CLINICAL TRIAL: NCT06286046
Title: A Phase 2, Open-label, Multicenter Study of Mitapivat in Subjects With Sickle Cell Disease and Nephropathy (RESIST)
Brief Title: A Study of Mitapivat in Participants With Sickle Cell Disease and Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG348-C-026; 2023-510289-28-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Nephropathy
Keywords: AG-348; Mitapivat
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases | interventions — mitapivat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mitapivat 100 mg (Experimental): Participants will receive mitapivat 100 milligrams (mg) tablet, orally, twice daily (BID) for up to 24 months.
  Interventions: Drug: Mitapivat

INTERVENTIONS:
Drug: Mitapivat — Tablets
  Other Names: AG-348; Mitapivat sulfate; AG-348 sulfate hydrate

SUMMARY:
The primary purpose of this study is to evaluate the effect of mitapivat on albumin creatinine ratio (ACR) response in participants with sickle cell disease (SCD) and nephropathy.

ELIGIBILITY:
Key Inclusion Criteria:

* Age of 16 years or older (except in France where participants must be aged 18 years or older);

  * Females must be post-menarche;
* Documented diagnosis of sickle cell disease (Homozygosity for hemoglobin S [HbSS] or Hemoglobin S/Beta 0 [HbS/β0]-thalassemia);
* Hemoglobin concentration ≥ 5.5 and ≤ 10.5 grams per deciliter (g/dL) during the Screening Period. If more than one measurement is collected during the Screening Period, the average must be ≥ 5.5 and ≤ 10.5 g/dL;
* If taking hydroxyurea, the dose of hydroxyurea must have been stable for at least 90 days before Study Day 1 with no planned dose adjustment during the study and no sign of hematologic toxicity;

  * Discontinuation of hydroxyurea requires a 90-day washout before providing informed consent/assent;
* Two urine ACR results collected during the Screening Period, both of which must be ≥ 100 and < 2000 milligrams per gram (mg/g). One ACR result can be from an untimed urine sample collected as part of a clinic visit. The other ACR result must be from a urine sample that is the first (or second) morning void on another day;
* One ACR result > 100 mg/g within 24 weeks before providing informed consent/assent;
* If taking Angiotensin-converting enzyme (ACE) inhibitor or Angiotensin receptor blockers (ARB) therapy, must have been on stable dose for at least 90 days before providing informed consent/assent with no planned dose adjustment during the study;
* Women of childbearing potential (WOCBP) must be abstinent of sexual activities that may induce pregnancy as part of their usual lifestyle or agree to use 2 forms of contraception, one of which must be considered highly effective, from the time of providing informed consent/assent, throughout the study, and for 28 days after the last dose of study drug. The second form of contraception can include an acceptable barrier method.

Key Exclusion Criteria:

* Pregnant, breastfeeding, or parturient;
* Currently receiving regularly scheduled red RBC transfusion therapy (also termed chronic, prophylactic, or preventative transfusion); episodic transfusion in response to worsened anemia or vaso-occlusive crisis (VOC) is permitted;
* Have received an RBC transfusion within 60 days before providing informed consent/assent or during the Screening Period;
* Hospitalized within 14 days before providing informed consent/assent or during the Screening Period either for a sickle cell disease pain crisis (SCPC) or other vaso-occlusive event;
* More than 10 SCPCs in the 52 weeks before providing informed consent/assent;
* History of stroke or meeting criteria for primary stroke prophylaxis (history of 2 transcranial Doppler [TCD] measurements ≥ 200 centimeters per second (cm/s) by nonimaging TCD or ≥ 185 cm/s by imaging TCD) at any time;
* Renal dysfunction as defined by an eGFR < 45 milliliters per minute (mL/min)/1.73 meters per square (m^2) by the Chronic Kidney Disease Epidemiology Collaboration creatinine equation (National Kidney Foundation, 2021b) at Screening;
* History of renal disease due to another disorder (e.g., diabetes, hypertension, primary focal segmental glomerulosclerosis, autoimmune) unrelated to SCD at any time;
* Evidence of acute kidney injury (in the opinion of the Investigator) within 4 weeks before informed consent/assent or during Screening Period.
* Currently undergoing renal replacement therapy (i.e., hemodialysis, peritoneal dialysis, hemofiltration, kidney transplantation);
* History of kidney transplant at any time;
* Currently receiving treatment with a disease-modifying therapy for SCD (eg, voxelotor, crizanlizumab, L-glutamine), except for hydroxyurea. The last dose of such therapies must have been administered at least 90 days before starting study drug;
* Currently receiving treatment with hematopoietic stimulating agents; the last dose must have been administered at least 90 days before starting study drug;

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Albumin Creatinine Ratio (ACR) Response | Baseline up to 6 months
  The ACR response is defined as a decrease of 30% or more in ACR from the baseline to Month 6.

SECONDARY OUTCOMES:
Change From Baseline in Cystatin C and Creatinine-based Estimated Glomerular Filtration Rate (eGFRcr-cys) | Baseline up to 25 months
Change From Baseline in Albumin Creatinine Ratio (ACR) | Baseline up to 25 months
Percentage of Participants With Stable ACR | Baseline up to 6 months
  Stable ACR is defined as Month 6 ACR within 20% of baseline ACR.
Annualized Rate of Emergency Room (ER) Visits | Up to 24 months
Annualized Rate of Days of Hospitalizations | Up to 24 months
Type, Frequency, Severity, and Relationship to Study Drug of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbasi M, Srivastava A, Saraf SL. Management of Kidney Disease with Sickle Cell Disease. J Am Soc Nephrol. 2025 Oct 1;36(10):2041-2054. doi: 10.1681/ASN.0000000804. Epub 2025 Jun 26. PMID 40569673